CLINICAL TRIAL: NCT01019135
Title: A Randomized Controlled Trial of Women's Adherence to Women-only, Home-based and Traditional Cardiac Rehabilitation (Cardiac Rehabilitation for Her Heart Event Recovery [CR4HER])
Brief Title: Cardiac Rehabilitation for Heart Event Recovery (HER)
Acronym: CR4HER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Sherry Grace, Director of Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Cardiac Rehab for Women
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Ischemia; Acute Coronary Syndrome; Heart Disease; Coronary Artery Disease
Keywords: Women; Cardiac Care Facilities; Patient satisfaction; Patient participation; Patient compliance; Randomized Control Trial; Coronary artery bypass; Angioplasty, transluminal, percutaneous coronary
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome; Heart Diseases; Coronary Artery Disease; Patient Satisfaction; Patient Participation; Patient Compliance | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Women-Only Cardiac Rehabilitation (Active Comparator): The women-only CR programs include on-site group exercise training sessions 1-2 days/week. Participants are encouraged to walk at home on alternate days of the week. Education sessions are also given in a group format, wherein participants engage in on-site female-only group exercise sessions, as well as female-only group education sessions.
  Interventions: Behavioral: Cardiac Rehabilitation
- Co-ed Cardiac Rehabilitation (Active Comparator): The traditional hospital-based co-ed CR programs include on-site group exercise training sessions 1-2 days/week. Participants are encouraged to walk at home on alternate days of the week. Education sessions are also given in a group format.
  Interventions: Behavioral: Cardiac Rehabilitation
- Home-Based Cardiac Rehabilitation (Active Comparator): In the monitored home-based programs, patients attend an intake appointment where an exercise test is performed as the basis for exercise prescription. Patients are given written guidelines for aerobic conditioning based on their treadmill test. Patients are cautioned about symptoms, and taught how to check their heart rate during walking sessions. Patients are provided with reading materials regarding CVD, risk factors and lifestyle modification. These are discussed with an allied health professional from the home-based CR program by telephone during weekly scheduled telephone calls.
  Interventions: Behavioral: Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — comparison of multiple cardiac rehabilitation program models

SUMMARY:
The purpose of this study is to compare women's cardiac rehabilitation program adherence across three program models.

DETAILED DESCRIPTION:
Heart disease is the leading cause of morbidity and mortality for women in Canada. Cardiac rehabilitation (CR) is an outpatient secondary prevention program composed of structured exercise and comprehensive education and counseling. CR participation results in lower morbidity and mortality, among other benefits. Unfortunately, women are significantly less likely to adhere to these programs than men. While the traditional model of CR care is a hospital-based mixed-sex program, women are the minority in such programs, and state that these programs do not meet their care preferences. Two other models of CR care have been developed: hospital-based women-only (sex-specific) and monitored home-based programs. Other than through our controlled pilot testing of 36 patients, women's adherence to these program models is not well known.

CR4HER is a 3 parallel arm pragmatic RCT designed to compare program adherence to traditional hospital-based CR with males and females, home-based CR, and women-only hospital-based CR. Power calculations based on our pilot study suggest a sample size of 261 patients is needed to detect a difference in adherence by program model using ANCOVA. Participants are female CAD, acute coronary syndrome, percutaneous coronary intervention, bypass surgery, or valve surgery inpatients recruited from 5 hospitals. Also, female patients referred to participating cardiac rehabilitation (3) centres with one of the aforementioned diagnosis will be approached to participate. The primary outcome variable is program adherence operationalized as CR site-reported percentage of prescribed sessions completed by phone or on-site, as reported by a staff member who is blind to study objectives. Secondary outcomes are exercise capacity operationalized as VO2peak on a graded stress test, and exercise, dietary, smoking and medication adherence behaviours measured in hospital and 1 week post-CR. By identifying the CR program model which results in the greatest adherence for women, we can optimize their participation and potentially their cardiac outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Documented coronary artery disease and/or acute coronary syndrome diagnosis and/or revascularization (coronary bypass graft or angioplasty) and/or valve surgery
* Work or reside in Greater Toronto Area
* Proficiency in English language
* Written approval to participate in CR by the patient's cardiac specialist or general practitioner
* Eligible for home-based CR

Exclusion Criteria:

* musculoskeletal, neuromuscular, visual, cognitive or non-dysphoric psychiatric condition, or any serious or terminal illness not otherwise specified which would preclude CR eligibility based on CR guidelines
* physician deems patient not suitable for CR at time of intake exercise stress test
* planning to leave the area prior to the anticipated end of participation
* being discharged to a long-term care facility
* participation in another clinical trial with behavioral interventions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L Grace, PhD, Principal Investigator — University Health Network & York University; Heather M Arthur, PhD, Study Chair — McMaster University; Paul Oh, MD, Study Chair — Toronto Rehabilitation Institute; Caroline Chessex, MD, Study Chair — University Health Network, Toronto; Stephanie Brister, MD, Study Chair — University Health Network, Toronto
Locations (5):
- Canada (5):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Mount Sinai, Toronto, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Grace SL, Midence L, Oh P, Brister S, Chessex C, Stewart DE, Arthur HM. Cardiac Rehabilitation Program Adherence and Functional Capacity Among Women: A Randomized Controlled Trial. Mayo Clin Proc. 2016 Feb;91(2):140-8. doi: 10.1016/j.mayocp.2015.10.021. Epub 2015 Dec 10. PMID 26682921

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Started | 55 | 59 | 55
Completed | 35 | 40 | 24
Not Completed | 20 | 19 | 31
Not completed — Did not receive allocated intervention | 12 | 6 | 25
Not completed — Did not attend CR | 8 | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation | Total
Number analyzed (Participants) | 55 | 59 | 55 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.22 (10.21) | 61.56 (9.73) | 63.13 (10.94) | 63.64 (10.42)
Sex/Gender, Customized [Number; unit: participants]
  Females | 55 | 59 | 55 | 169
Race/Ethnicity, Customized [Number; unit: participants]
  White | 26 | 32 | 32 | 90
  Other | 29 | 27 | 23 | 79
Region of Enrollment [Number; unit: participants]
  Canada | 55 | 59 | 55 | 169

OUTCOME MEASURES:

1. Primary Outcome: CR Program Adherence
Time Frame: 6 months
Population: Participants with available data for adherence
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 54 | 53 | 46
percentage of sessions attended | 54.40 (34.72) | 51.33 (35.7) | 58.12 (35.39)

2. Secondary Outcome: Exercise Capacity
Description: Exercise capacity as measured by VO2peak on a graded stress test.
Time Frame: 6 months
Population: Participants with available data for exercise capacity
Measure: Mean (Standard Deviation); unit: mL/(kg·min)
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 28 | 30 | 32
mL/(kg·min) | 21.6071 (7.18327) | 20.8450 (6.51039) | 21.0734 (8.99184)

3. Secondary Outcome: Exercise
Description: Mean daily steps as measured by a pedometer over 7 days
Time Frame: 6 months
Population: Participants with available data for exercise
Measure: Mean (Standard Deviation); unit: Daily steps
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 21 | 15 | 19
Daily steps | 5296.9660 (2803.16268) | 6129.7143 (3107.17927) | 6694.3308 (4463.47290)

4. Secondary Outcome: Self-reported Exercise
Description: The Godin Leisure-time Exercise Questionnaire will be administered in the pre and post-test surveys. It is a brief and reliable instrument to assess usual leisure-time physical activity behaviour during a one-week period. For the first question, weekly frequencies of strenuous, moderate, and light activities are multiplied by nine, five, and three, respectively. Part two of the questionnaire calculates the frequency of weekly leisure-time activities pursued. Total weekly leisure activity is calculated by summing the products of the separate components. Scores begin at zero, with higher scores indicating greater physical activity. For example, scores equal to or greater than 20 are indicative of someone who is "active". There is no max score.
Time Frame: 6 months
Population: Participants with available data for self-reported exercise
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 37 | 40 | 31
Scores on a scale | 31.3243 (23.46517) | 31.4 (21.7922) | 29.5645 (14.29612)

5. Secondary Outcome: Diet
Description: The Diet Habit Survey was used to assess diet. It is an inexpensive, reliable, and valid instrument for rapid assessment of eating habits and diet composition. Its 9 questions are related to the consumption of cholesterol, saturated fat, complex carbohydrate (including fiber), and salt.
  Greater scores indicate better diets, both for the total score and for each area. The total score indicates the level of fat in the diet (with scores equal to or greater than 236 corresponding to a low-fat diet 20% or less). Scores can begin at 56 and have no upper range.
Time Frame: 6 months
Population: Participants with available data for diet
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 38 | 41 | 36
Scores on a scale | 202.2019 (24.34676) | 202.3477 (27.54240) | 213.9834 (32.89330)

6. Secondary Outcome: Medication Adherence
Description: The 4-item Morisky Medication Adherence Scale was used, which is scored as yes = 0, no = 1, such that a higher score indicates higher medication adherence. Scores range from 0 to 4, with patients scoring 2 or above considered adherent.
Time Frame: 6 months
Population: Participants with available data for medication adherence
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 38 | 42 | 36
Scores on a scale | 3.6842 (0.57447) | 3.5238 (0.80359) | 3.5833 (0.76997)

7. Secondary Outcome: Smoking
Description: Current smoking status
Time Frame: 6 months
Population: Participants with available data for current smoking status. Reported values in the table represent number of participants who were current smokers.
Measure: Number; unit: Participants
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Number analyzed (Participants) | 38 | 42 | 36
Participants | 1 | 3 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Women-Only Cardiac Rehabilitation | Co-ed Cardiac Rehabilitation | Home-Based Cardiac Rehabilitation
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/59 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/59 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No